CLINICAL TRIAL: NCT03093545
Title: Effect of Rabies Immunoglobulin on Immunogenicity of Post-exposure Rabies Vaccination in Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: VINS Bioproducts Ltd. (Unknown); Biogentech Co.,LTD (Unknown)
Responsible Party: Principal Investigator, Jatuporn Sirikun, Principal Investigator, Mahidol University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Si178/2015
Record Dates: First submitted 2017-01-24; First posted 2017-03-28 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Rabies
Keywords: rabies; obese; immunoglobulin; rabies vaccine; post-exposure; immunogenicity
MeSH Terms: conditions — Rabies; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal BMI or underweight (< 24 Kg/m2) (Other)
  Interventions: Biological: Equine Rabies Immunoglobulin; Biological: Purified chick-embryo cell rabies vaccine
- Obese (BMI > 30 Kg/m2) (Experimental)
  Interventions: Biological: Equine Rabies Immunoglobulin; Biological: Purified chick-embryo cell rabies vaccine

INTERVENTIONS:
Biological: Equine Rabies Immunoglobulin — 40 IU per kg of body weight of ERIG at Day 0
  Other Names: ERIG
Biological: Purified chick-embryo cell rabies vaccine — 1 ml of PCEC Rabies vaccine on days 0, 3, 7, 14 and 28.
  Other Names: PCEC

SUMMARY:
A single center, prospective cohort, open-label study of rabies post exposure program with equine rabies immunoglobulin (ERIG) and purified chick-embryo cell (PCEC) rabies vaccine in WHO category III exposed patients at Siriraj Hospital, Thailand aims to compare serum RVNA responses between obese (BMI > 30 kg/m2) and normal weight/underweight (BMI < 25 kg/m2) and to evaluate adverse events occurring after immunization on days 7, 14 and 28.

DETAILED DESCRIPTION:
A single center, prospective cohort, open-label study of rabies post exposure program with equine rabies immunoglobulin (ERIG) and purified chick-embryo cell (PCEC) rabies vaccine in WHO category III exposed patients at Siriraj Hospital, Thailand aims to compare serum RVNA responses between obese (BMI > 30 kg/m2) and normal weight/underweight (BMI < 25 kg/m2) and to evaluate adverse events occurring after immunization on days 7, 14 and 28.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ages of >= 18 years and older;
2. Experienced WHO category III rabies exposure excluding presenting wound at eye(s) or eye lid(s);
3. Either a) obese with BMI >= 30 or b) normal weight and/or underweight with BMI < 25;
4. Agree to independently consent to participate in all study procedures.

Exclusion Criteria:

1. Positive skin test to ERIG or known hypersensitivity to ERIG or its excipients;
2. Co-enrolment with other studies or participated in other investigational drug studies or use of other investigational drugs within 4 weeks or five times the half-life of the investigational drug;
3. Female patients who are currently pregnant or breast feeding.
4. Presenting with wound at eye(s) or eye lid(s);
5. Receiving rabies vaccination more than 7 days for this exposure;
6. History of complete pre-exposure or post-exposure regimen with at least 3 doses;
7. Known of allergic to egg or poultry meat;
8. History of previous exposure to equine sera
9. Significant illness that might harm or increase the risk to the patients;
10. History of drug abuse or alcoholism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-03; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
The difference of rabies virus neutralizing antibody (RVNA) levels between obese and normal/underweight patients. | At day 7 prior to vaccination.
  To compare RVNA levels between obese and normal/underweight patients.
The difference of rabies virus neutralizing antibody (RVNA) levels between obese and normal/underweight patients. | At day 14 prior to vaccination.
  To compare RVNA levels between obese and normal/underweight patients.
The difference of rabies virus neutralizing antibody (RVNA) levels between obese and normal/underweight patients. | At day 28 prior to vaccination.
  To compare RVNA levels between obese and normal/underweight patients.

SECONDARY OUTCOMES:
Incidence of adverse event | From day 0 to day 60
  Number of participants with ERIG or PCEC-related adverse events as assessed by investigator as per CTCAE v4.03.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Siriraj Hospital, Mahidol University, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
No plan to provide individual participant data (IPD). However, other researcher could request IPD from principal investigator.